CLINICAL TRIAL: NCT00682162
Title: Impact of Acupuncture on Vasomotor Rhinitis: a Randomised Placebo Controlled Pilot Study
Brief Title: Impact of Acupuncture on Vasomotor Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: PD Dr. Dominik Irnich, Multidisciplinary Pain Centre, Department of Anaesthesiology, University of Munich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPC-UM-0001-DI
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2008-05

CONDITIONS: Vasomotor Rhinitis; Acupuncture
Keywords: acupuncture; randomised controlled trial; placebo; sham laser; vasomotor rhinitis
MeSH Terms: conditions — Rhinitis, Vasomotor | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham-laser acupuncture (Sham Comparator): The sham-laser acupuncture treatment consisted of 5 sessions, all patients completed a recovery time after treatment of 30 min duration. The sessions were administered over a period of 5 weeks (one session per week). Sham-laser acupuncture was applied at the same points as the acupuncture treatment. A deactivated laser pen (Seirin, 3B Scientific GmbH, Hamburg, Germany) that could only beam normal red light rather than laser was used. The total number of acupuncture points utilized was equal to the acupuncture group. Every point was treated for 30 sec with the total treatment time of 20 minutes.
  Interventions: Device: Sham-laser acupuncture
- Acupuncture (Active Comparator): The treatment consisted of 5 sessions, all patients completed a recovery time after treatment of 30 min duration. The sessions were administered over a period of 5 weeks (one session per week). The acupuncture treatment was semi-standardised. It consisted of a basic pool of 6 body acupuncture points. Five additional acupuncture body points together with auricular points formed an individual pool. After needle insertion, the needle was manipulated until the subject obtained the de-Qi response (a deep aching or full feeling at the needle, [22]). After obtaining the de-Qi response, there was no further manipulation of the needle. Each session lasted 20 minutes.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — The treatment consisted of 5 sessions, all patients completed a recovery time after treatment of 30 min duration. The sessions were administered over a period of 5 weeks (one session per week). The acupuncture treatment was semi-standardised. It consisted of a basic pool of 6 body acupuncture points. Five additional acupuncture body points together with auricular points formed an individual pool. After needle insertion, the needle was manipulated until the subject obtained the de-Qi response (a deep aching or full feeling at the needle, [22]). After obtaining the de-Qi response, there was no further manipulation of the needle. Each session lasted 20 minutes.
  Arms: Acupuncture
Device: Sham-laser acupuncture — The sham-laser acupuncture treatment consisted of 5 sessions, all patients completed a recovery time after treatment of 30 min duration. The sessions were administered over a period of 5 weeks (one session per week). Sham-laser acupuncture was applied at the same points as the acupuncture treatment. A deactivated laser pen (Seirin, 3B Scientific GmbH, Hamburg, Germany) that could only beam normal red light rather than laser was used. The total number of acupuncture points utilized was equal to the acupuncture group. Every point was treated for 30 sec with the total treatment time of 20 minutes.
  Arms: Sham-laser acupuncture

SUMMARY:
Chronic rhinitis without an allergic or infectious aetiology (vasomotor rhinitis) is a common disease for which there are only poor therapeutic treatment options. The current placebo controlled partially double blinded pilot study evaluated the effects of acupuncture on the symptoms of vasomotor rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* term of sickness > 3 month
* negative allergic testing

Exclusion Criteria:

* term of sickness < 3 month
* previous nasal surgeries
* polyposis nasi
* contraindications regarding acupuncture (such as: risk of bleeding, pregnancy)
* psychologic disorders
* drug addiction
* autoimmune disease
* other severe disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1998-01; Primary Completion 1999-01 (Actual); Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
The main outcome measure was the alteration of the nasal sickness score (NSS; scoremax 27). | 5 weeks

SECONDARY OUTCOMES:
Secondary outcome measures were the evaluation of a subjective symptoms score by patients' diaries and of their quality of life (SF-12 health survey). | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Irnich, PD. Dr., Principal Investigator — Multidisciplinary Pain Centre, Department of Anaesthesiology, University of Munich, Germany
Locations (2):
- Germany (2):
  - Department of otorhinolaryngology of the University of Munich, Munich
  - Multidisciplinary Pain Centre, Department of Anaesthesiology, University of Munich,, Munich

REFERENCES:
- [Result] Fleckenstein J, Raab C, Gleditsch J, Ostertag P, Rasp G, Stor W, Irnich D. Impact of acupuncture on vasomotor rhinitis: a randomized placebo-controlled pilot study. J Altern Complement Med. 2009 Apr;15(4):391-8. doi: 10.1089/acm.2008.0471. PMID 19388861